CLINICAL TRIAL: NCT04636229
Title: A Phase 3 Prospective, Multicenter, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy of Amniotic Suspension Allograft (ASA) in Patients With Osteoarthritis of the Knee
Brief Title: Efficacy of Amniotic Suspension Allograft in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organogenesis (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19 OA 001 ASA
Record Dates: First submitted 2020-11-05; First posted 2020-11-19 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Knee; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, randomized, double-blind, placebo-controlled study of ASA in patients with OA of the knee. Patients will be randomly assigned in a 1:1 ratio to receive a single IA injection of 2 mL of ASA (plus 2 mL of normal saline) or 4 mL of normal saline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All clinic staff who may be involved in making assessments of safety will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ASA (Experimental): Participants receive a single IA injection of 2 mL of ASA (plus 2 mL of normal saline)
  Interventions: Biological: Amniotic Suspension Allograft
- Placebo (Placebo Comparator): Participants receive a single IA injection of 4 mL of normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Amniotic Suspension Allograft — This investigational product is a cryopreserved product derived from human amnion and cells from the amniotic fluid.
  Arms: ASA
Drug: Placebo — Matching placebo is 0.9% normal saline: 4 mL to be injected IA.
  Arms: Placebo

SUMMARY:
This study is being conducted to evaluate the efficacy and safety of ASA compared to placebo in the management of osteoarthritis (OA) symptoms of the knee.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, double-blind, placebo-controlled Phase 3 study of ASA in patients with OA of the knee. Initially, 474 subjects are planned for inclusion in this study using a group sequential design with two interim analyses and a final analysis. Sample size re-estimation is planned at the second interim analysis. Based on conditional power, the maximum sample size may be increased to up to 700 patients. Patients will be randomly assigned in a 1:1 ratio to receive a single intra-articular (IA) injection of 2 mL of ASA (plus 2 mL of normal saline) or 4 mL of normal saline.

Patients will be screened after informed consent is obtained. Eligible patients will be randomized to receive a single IA injection on Day 1. They will have serial assessments of knee pain, function, and symptoms scores, as well as safety assessments for up to 52 weeks after administration of the study drug.

The planned sequence and maximum duration of the study periods will be as follows:

* Screening: 2 weeks
* Treatment: 1 day
* Follow-up: 52 weeks

The maximum treatment duration for each patient is 1 day.

The maximum study duration for each patient is 54 weeks.

Efficacy will be assessed via Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and Outcome Measures in Rheumatology-Osteoarthritis Research Society International (OMERACT-OARSI) responder rates.

Safety will be assessed via monitoring of adverse events (AEs), safety laboratory testing, vital signs, physical examination, and concomitant medication use.

An independent data monitoring committee (DMC) with a defined charter will review study data and make preliminary decisions relative to interim analyses.

The assessments that are used in this study are standard, and are generally recognized as reliable, accurate, and relevant.

No pediatric patients will be included as OA of the knee is an age-related disorder and rarely occurs in patients under the age of 18 years. The sponsor plans to submit a waiver for studies in all pediatric age subgroups.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 18 years of age or older
2. Diagnosis of OA of the knee by a combination of clinical and radiographic findings
3. OA of the knee with Kellgren and Lawrence radiographic classification (Grade 2-4 inclusive) confirmed by posterior-anterior, weight-bearing, fixed flexion radiography with 10° caudal beam angulation. A specially designed positioning frame will be used to standardize the positioning for image acquisition.
4. Patients who have failed to adequately respond for at least 6 months to at least 2 OA therapies that include conservative, non-pharmacological therapy and simple analgesics (e.g., acetaminophen); nonsteroidal anti-inflammatory drugs (NSAIDS); avoidance of activities that cause joint pain; exercise; weight loss; physical therapy; and removal of excess fluid from the knee
5. Overall pain score over the previous 7 days of 11 or more on the WOMAC Pain scale.
6. Body mass index (BMI) < 40 kg/m²
7. If female, must be postmenopausal (for at least 2 years), surgically sterilized (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), sexually abstinent, or willing and able to use 2 methods of contraception from Day 1 through 12 months after treatment
8. Males who are not surgically sterile (vasectomy) for at least 6 months prior to screening must confirm their willingness to use adequate methods of contraception from Day 1 through 12 months after treatment
9. Willing to agree not to use illicit drugs during the study, and to have illicit drug testing at screening and at later time points, if illicit drug use is suspected during the study
10. Able to comply with study requirements and complete the full sequence of protocol-related procedures and evaluations, including post-hospitalization, out-patient, and follow-up visits
11. Able to understand and provide written informed consent

Exclusion Criteria:

1. Use of pain medication (including NSAIDs and cannabidiol [CBD] oil) less than 15 days before treatment (acetaminophen allowed)
2. Regular use of anticoagulants
3. Symptoms of locking, intermittent block to range of motion, or loose body sensation that could indicate meniscal displacement or an IA loose body
4. Corticosteroid injection into the index knee within 3 months prior to screening
5. Viscosupplement (e.g., hyaluronic acid [HA]) injection, platelet-rich plasma injection, bone marrow aspirate (BMA) or bone marrow aspiration concentrate (BMAC), placental-derived tissue/cells, adipose tissue, or any other autologous or allogeneic product into the index knee within 6 months prior to screening
6. Patients with known hypersensitivity reactions to ASA or any of its constituents (e.g., HA, dimethyl sulfoxide [DMSO])
7. Knee surgery on the index knee within 12 months prior to screening and/or planned knee surgery during the study
8. Knee surgery on the contralateral knee within 6 months prior to screening and/or planned knee surgery during the study
9. Acute index knee trauma within 3 months prior to screening
10. Knee effusion requiring aspiration of the index or contralateral knee within 3 months prior to screening
11. Contralateral knee pain ≥ 4 on the WOMAC Pain scale on most days during the past week.
12. Current therapy with any immunosuppressive therapy, including corticosteroids (> 5 mg/day of prednisone)
13. Clinically significant findings on the screening laboratory tests or physical examination that are not specific to OA of the knee and may interfere with study conduct or interpretation of data or increase patient risk
14. Clinically significant intercurrent illness, medical condition, non-knee pain, or medical history (including neurological or mental illness, human immunodeficiency virus, fibromyalgia, complex regional pain syndrome, or any active infection, including hepatitis B or C) that could jeopardize the patient safety, limit participation, or compromise interpretation of data derived from the patient
15. Active alcohol or substance use disorder, or any other reason that would make it unlikely for the patient to comply with study procedures
16. Females who are pregnant (positive pregnancy test at screening or prior to treatment) or lactating
17. Participation in another clinical trial within the 30 days (or 5 half-lives of the investigational compound, whichever is longer) before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
The difference in change from baseline in WOMAC Pain scale at 6 months between ASA- and placebo-treated patients | Baseline to Week 26
  The Western Ontario and McMaster Universities (WOMAC®) Osteoarthritis Index is a questionnaire that measures pain, stiffness, and function both independently and collectively, using a Likert 3.1, 5-point scale. The Likert Scale uses the following descriptors for all items: none, mild moderate, severe, and extreme, corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.

SECONDARY OUTCOMES:
The difference between changes from baseline for ASA- and placebo- treated patients in WOMAC Function at 6 months | Baseline to Week 26
  The Western Ontario and McMaster Universities (WOMAC®) Osteoarthritis Index is a questionnaire that measures pain, stiffness, and function both independently and collectively, using a Likert 3.1, 5-point scale. The Likert Scale uses the following descriptors for all items: none, mild moderate, severe, and extreme, corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
The difference between changes from baseline for ASA- and placebo-treated patients in the OMERACT-OARSI responder rate at 6 months | Baseline to Week 26
  Outcome Measures in Rheumatoid Arthritis Clinical Trials - Osteoarthritis Research Society International. (OMERACT-OARSI) Responders are defined as participants with high improvement in pain or function.
The difference between changes from baseline for ASA- and placebo-treated patients in WOMAC Pain at 3 months | Baseline to Week 12
  The Western Ontario and McMaster Universities (WOMAC®) Osteoarthritis Index is a questionnaire that measures pain, stiffness, and function both independently and collectively, using a Likert 3.1, 5-point scale. The Likert Scale uses the following descriptors for all items: none, mild moderate, severe, and extreme, corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
The difference between changes from baseline for ASA- and placebo- treated patients in non-inferiority of WOMAC Function at 3 months | Baseline to Week 12
  The Western Ontario and McMaster Universities (WOMAC®) Osteoarthritis Index is a questionnaire that measures pain, stiffness, and function both independently and collectively, using a Likert 3.1, 5-point scale. The Likert Scale uses the following descriptors for all items: none, mild moderate, severe, and extreme, corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
The difference between changes from baseline for ASA- and placebo-treated patients in the OMERACT-OARSI responder rate at 3 months | Baseline to Week 12
  Outcome Measures in Rheumatoid Arthritis Clinical Trials - Osteoarthritis Research Society International. (OMERACT-OARSI) Responders are defined as participants with high improvement in pain or function.
The difference between changes from baseline for ASA- and placebo-treated patients in the WOMAC Total at 6 months | Baseline to Week 26
  The Western Ontario and McMaster Universities (WOMAC®) Osteoarthritis Index is a questionnaire that measures pain, stiffness, and function both independently and collectively, using a Likert 3.1, 5-point scale. The Likert Scale uses the following descriptors for all items: none, mild moderate, severe, and extreme, corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
The difference between ASA- and placebo-treated patients in the WOMAC Stiffness at 6 months | Baseline to Week 26
  The Western Ontario and McMaster Universities (WOMAC®) Osteoarthritis Index is a questionnaire that measures pain, stiffness, and function both independently and collectively, using a Likert 3.1, 5-point scale. The Likert Scale uses the following descriptors for all items: none, mild moderate, severe, and extreme, corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
The difference between changes from baseline for ASA- and placebo- treated patients in the WOMAC Total at 3 months | Baseline to Week 12
  The Western Ontario and McMaster Universities (WOMAC®) Osteoarthritis Index is a questionnaire that measures pain, stiffness, and function both independently and collectively, using a Likert 3.1, 5-point scale. The Likert Scale uses the following descriptors for all items: none, mild moderate, severe, and extreme, corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
The difference between changes from baseline for ASA- and placebo-treated patients in the WOMAC Stiffness at 3 months | Baseline to Week 12
  The Western Ontario and McMaster Universities (WOMAC®) Osteoarthritis Index is a questionnaire that measures pain, stiffness, and function both independently and collectively, using a Likert 3.1, 5-point scale. The Likert Scale uses the following descriptors for all items: none, mild moderate, severe, and extreme, corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Incidence of adverse events (AEs) | Baseline to Week 52
  An AE is any untoward medical occurrence in a clinical study patient administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product.
  This includes any occurrence that is new in onset or aggravated in severity or frequency from the baseline condition, or abnormal result of diagnostic procedures, including clinical laboratory test abnormalities.

CONTACTS AND LOCATIONS:
Locations (38):
- United States (38):
  - Central Research Associates, Birmingham, Alabama
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - AMR Mobile, Mobile, Alabama
  - Arizona Arthritis & Rheumatology Research, Glendale, Arizona
  - Fiel Family & Sports Medicine/ CCT Research, Tempe, Arizona
  - Arizona Arthritis & Rheumatology Research, Tucson, Arizona
  - Tri West Research Associates, El Cajon, California
  - Horizon Clinical Research Center, La Mesa, California
  - Actca, A Member of the Allliance Inc., Los Angeles, California
  - University of California at Los Angeles, Los Angeles, California
  - Stanford Medicine, Redwood City, California
  - University of California at Davis, Sacramento, California
  - AARDS Research, Inc., Aventura, Florida
  - Gulfcoast Research Institute, Sarasota, Florida
  - Pinnacle Trials, Inc., Stockbridge, Georgia
  - Injury Care Research, Boise, Idaho
  - Chicago Clinical Research Institute Inc, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Affinity Health, Oak Brook, Illinois
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Klein & Associates, MD, PA, Hagerstown, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Methodist Physicians Clinic/ CCT Researc, Fremont, Nebraska
  - Physician Research Collaboration, Lincoln, Nebraska
  - NYU Langone Health, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Lenox Hill Hospital (Northwell Health), New York, New York
  - M3 Emerging Medical Research, LLC, Durham, North Carolina
  - Moore Orthopedics and Sports Medicine, Morehead City, North Carolina
  - M3 Emerging Medical Research, LLC, Raleigh, North Carolina
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - University Orthopedics Center, Altoona, Pennsylvania
  - University Orthopedic Center, State College, Pennsylvania
  - PCPMG Clinical Research Unit, LLC, Greenville, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Affinity Health, Nashville, Tennessee
  - Cedar Health Research, LLC, Burleson, Texas
  - Spectrum Medical, Inc, Danville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Farr J, et al. A randomized controlled single-blind study demonstrating superiority of ASA injection over hyaluronic acid and saline control for modification of knee OA symptoms. J Knee Surg. 2019; https://doi.org/10.1055/s-0039-1696672. — https://pubmed.ncbi.nlm.nih.gov/31533151/